CLINICAL TRIAL: NCT02369640
Title: Learning From Errors During Simulation-based Ultrasound Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Martin G. Tolsgaard, MD, ph.d., postdoc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H-4-2015-FSP
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Simulation-based Ultrasound Training, Error-management Training, Training With Errors, Skills Transfer

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Error-avoidance training (Experimental): Study group 1: Error-avoidance training (Focusing on achieving the highest possible metrics score by avoiding errors).
  Interventions: Procedure: Error-management training vs error-avoidance training. Defined by training instructions.
- Error-management training (Experimental): Study group 2: Error-management training (Focusing on making errors and thinking of them in a positive way).
  Interventions: Procedure: Error-management training vs error-avoidance training. Defined by training instructions.

INTERVENTIONS:
Procedure: Error-management training vs error-avoidance training. Defined by training instructions. — . Error-avoidance training: The participants are instructed to follow the simulator program step-by-step, to achieve the highest possible simulator metric scores by making as few errors as possible, and only to follow the task required in the training program.
  Study group 2. Error-management training: The participants are required to complete the same training program as study group 1. The participants are instructed to experiment and explore on their own and to deliberately make errors during the task that they are instructed to perform. Participants are instructed to reflect on their errors based on the simulator metrics that they do not pass. Errors are framed as positive events and instructor comments may include statements such as "the more errors you make, the more you learn!" or "you have made an error? Great! Because now you can learn something new!"

SUMMARY:
During the past decades, simulation-based training has become essential for making trainees fit for clinical practice. Traditionally, trainees are instructed to practice with as few errors as possible during simulation-based training. However, recent evidence from the field of psychology suggests that transfer of learning may improve if trainees are encouraged to commit errors during training. The aim of this study is to assess on performances with real patients the effect of error-management instructions compared to error-avoidance instructions during simulation-based virtual reality ultrasound training.

This study is planned as a randomized controlled trial. Participants include medical students with no prior simulation practice at the fifth or sixth year of medical school. All participants receive 3 hours simulation-based ultrasound training focusing on fetal weight estimation. The participants (N=60) are randomized into two groups: Participants in group 1 are instructed to follow the simulator program step-by-step to achieve the highest possible simulator metric scores by making as few errors as possible. Participants in group 2 are instructed to experiment and explore and to deliberately make errors during training. A simulation-based pre- and post-test is administered before and after training.

Participants are scheduled to perform a transfer test seven to ten days after simulation training. The transfer test consists of fetal weight estimation on a real patient. The primary outcome is weight deviation of participant measurements compared to expert findings. Secondary outcomes include performance assessments of pre-, post- and transfer test performances by blinded ultrasound experts using the Objective Structured Assessment of Ultrasound Skills (OSAUS) scale. Using an alpha level of 0.05, an effect size of 0.80, and a power of 0.80, 25 participants are needed in the two study groups. Loss to follow-up of up to 20% of study participants is anticipated, resulting in 30 participants in each study group.

ELIGIBILITY:
Inclusion Criteria:

* are enrolled during the fifth or sixth year of medical school
* provide written informed consent

Exclusion Criteria:

* have clinical or simulator ultrasound experience

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy | 7-10 days later in a tranfer test
  The primary outcome is diagnostic accuracy during the transfer test performances. Diagnostic accuracy is determined as the percentage deviation from the fetal weight estimation performed by an experienced sonographer (i.e. an ultrasound expert).

SECONDARY OUTCOMES:
performance scores based on the Objective Structured Assessment of Ultrasound Skills (OSAUS) scale | 7-10 days in a tranfer test
  Secondary outcome measures include performance scores based on the Objective Structured Assessment of Ultrasound Skills (OSAUS) scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Juliane Marie Center, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Dept. of Fetal Medicine, Juliane Marie Centre, Copenhagen O